CLINICAL TRIAL: NCT02884453
Title: Proof-of-concept Study of Ibrutinib in c-MYC and HER2 Amplified Oesophagogastric Carcinoma
Acronym: iMYC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4449
Record Dates: First submitted 2016-07-21; First posted 2016-08-31 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Gastrooesophageal Cancer
Keywords: gastrooesophageal carcinoma
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ibrutinib (Experimental): ibrutinib delivered orally at a dose of 560mg once daily continuously on a 4 weekly cycle until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: ibrutinib

INTERVENTIONS:
Drug: ibrutinib — Ibrutinib (PCI-32765) is a first-in-class, potent, orally-administered, covalently-binding small molecule inhibitor of Bruton's tyrosine kinase (BTK) currently under development for the treatment of B-cell malignancies. Ibrutinib is being co-developed by Janssen Research & Development, LLC and Pharmacyclics Inc.
  Other Names: JNJ-54179060; IMBRUVICA; PCI-32765

SUMMARY:
Some cancers of the oesophagus and stomach express excessive copies of either the cMYC (Myelocytomatosis oncogene) gene, the HER2 (Human epidermal growth factor receptor 2) gene or both. These genes may potentially contribute to the growth and spread of cancer.Ibrutinib is a drug that is already used in the treatment of certain cancers of the immune system.

There is preclinical evidence that it shows activity against gastric and stomach cancer cells over-expressing cMYC and HER2 genes.

The iMYC study will assess the activity of ibrutinib in cancers of the oesophagus and stomach which over-express these genes and which have previously been treated with standard chemotherapies.

Any anti-cancer activity seen will be measured and correlated with metabolic changes on FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) - PET (positron emission tomography) scan, changes in DNA and circulating tumour cells in the blood, and molecular changes in the cancer itself through the use of optional repeat tumour biopsies. If an effect is seen it could provide justification for further research in this group of patients.

Patients will be eligible if they have advanced cancer of the oesophagus or stomach and have been treated with at least one line of prior therapy. The study will be conducted at the Royal Marsden Hospital at its Sutton and Chelsea sites.

It will involve an initial group of up to 17 patients. Screening, recruitment and follow up will last for 3 years in total.

Patients wishing to take part must consent to having their cancer biopsied to test for cMYC and HER2 amplification, as well as a number of imaging and blood tests. There are optional further tumour biopsies whilst on study.

Patients will be treated with ibrutinib until progression of their disease or unacceptable toxicity.

DETAILED DESCRIPTION:
This is an open-label, single-arm phase II study. Patients will receive standard dose single-agent ibrutinib delivered orally at a dose of 560mg once daily continuously on a 4 weekly cycle until disease progression or unacceptable toxicity occurs.

Single arm, open label means that both researchers and participants know the treatment which is being administered, and all participants in the trial will receive the study drug ibrutinib.

A Phase 2 study was chosen as more information about the efficacy and toxicity of this drug in this specific group of patients is needed prior to considering a larger phase 3 study.

Eligible patients are those with advanced unresectable or metastatic oesophagogastric adenocarcinoma or squamous cell carcinoma who have been treated with at least 1 prior chemotherapy for advanced or metastatic disease. In the case of HER2 positive tumours, previous treatment with chemotherapy with or without a HER2 targeted agent is allowed.

There will be a two step enrollment process:

1. Enrollment for prescreening to establish cMYC and HER2 status (which may occur during 1st line treatment or after progression on 1st line treatment)
2. Enrollment for randomisation and treatment The patient will first be given the prescreening participant information sheet (PIS) and informed consent form (ICF) that has been approved by the Ethics Committee. They will have the study explained to them and be given the opportunity to ask questions. If they agree to take part, they will be asked to sign the approved consent form, and they will keep a copy of the signed consent form.

   Prescreening If a participant agrees to take part in the prescreening for the study a previously obtained sample of their cancer (usually a diagnostic biopsy) will be taken out of storage and sent to the trial laboratory where the tissue will be tested for both cMYC and HER2 amplification. If there is no archival tumour sample available or if the existing tumour sample is of insufficient quality, the patient will be given the option to consent to a pre-screening biopsy to obtain a fresh sample.

   A blood test will be taken for plasma DNA analysis including circulating tumour cell number, c-MYC copy number variation (by digital droplet PCR) and blood-borne biomarkers. It can take up to 4 weeks to get these results which is why we will try to pre-screen patients to avoid delays in treatment. When the patient's disease progresses on 1st line treatment and if they are a suitable candidate for second line treatment their team will confirm if there are spaces available on study according to the the patients cMYC and HER2 status.

   If there are spaces available they will be given the main study PIS and ICF that has been approved by the Ethics Committee. They will have the study explained to them and be given the opportunity to ask questions. If they agree to take part, they will be asked to sign the approved consent form, and they will keep a copy of the signed consent form

   Screening

   If a participant agrees to take part in the main study, assessments will be made to make sure that he/she is eligible for the study. Some of these assessments may already have been done as part of the participant's standard of care, in which case, the results of those tests may be used. The assessments that will be done are described below:

   Disease status Tumour sample details, c-MYC and HER2 status if re-tested Medical/surgical history Pregnancy testing for female patients World Health Organisation (ECOG) performance status Physical examination to assess all conditions that are current and ongoing. Vital signs: height, weight, pulse, systolic blood pressure and diastolic blood pressure ECG Tumour biopsy* Tumour assessments (RECIST v1.1), consisting of either staging CT or MRI imaging FDG-PET scan* Concomitant medication. Adverse events Blood tests for clinical biochemistry and haematology Urinalysis Blood tests for DNA analysis including Circulating Tumor Cell (CTC) number, c-MYC copy number variation (by digital droplet PCR) and bloodborne biomarker analysis*

   *These procedures will only be carried out once all other criteria for trial entry are met.

   If the results of screening tests confirm that the patient can take part in the study they will be asked to return to the clinic to see their doctor for assessments as detailed below during the study treatment period.

   Study treatment period During the treatment period the patient will be seen regularly in clinic.The treatment is oral capsules given once per day every day in cycles lasting 28 days. Patients will be seen on day 1, 8 and 15 of the first cycle of treatment and then on day 1 of every cycle (every four weeks) for the remainder of the study duration. When they stop being treated within the study they will have a 30 day follow up visit and then be followed up every 8 weeks, although this contact can be over the telephone.

   Before each treatment cycle, the patient will be examined and have safety blood tests to make sure that it is safe to proceed with treatment as mentioned below. Patients will have different procedures done at different times during the study treatment period including:

   Measurement of resting blood pressure and pulse rate before every treatment (at all study visits).

   Physical examination at the beginning of each cycle (every four weeks). Documentation of any changes in the medication taken and whether the patient has had any problems or discomfort since the last visit (at all study visits).

   An ECG at baseline and on completion of study, and at any further timepoint if clinically indicated Blood samples to check haematology and clinical chemistry results (every 4 weeks or if clinically indicated) Blood samples for plasma DNA analysis including CTC number, c-MYC copy number variation (by ddPCR) and bloodborne biomarker analysis. These will be taken on cycle 1 day 15, cycle 3 day 1 and then every 8 weeks (alternate cycles).

   Blood samples to assess pharmacokinetics of ibrutinib on cycle 1 day 8 (predose, 2 hours, 6 hours post dose) and one further sample on cycle 1 day 15.

   Assessment of the status of disease using CT or MRI imaging at week 8 and then every 8 weeks.

   Assessment with PET CT scan at baseline, day 14 and week 8 to correlate with tumour response and genetic changes seen Health related quality of life questionaires for the patient to fill out at the beginning of each cycle (every 4 weeks)

   As mentioned above, a biopsy at the time of screening is mandatory for entry into the trial. As part of the trial further optional biopsies will be offered to the patient:

   at day 14 (in all patients on ibrutinib) at week 8 (on those patients responding to ibrutinib) on discontinuation of study treatment (on those patients who have progressed on ibrutinib)

   Treatment discontinuation visit:

   When the patient withdraws from the study or treatment is permanently discontinued, they will need to attend the clinic for a visit and the following assessments will be carried out:

   Changes in the medication taken and any problems or discomfort since their last visit will be documented.

   If the patient has a side effect at their final study visit or withdrawal visit then the study doctor may wish to contact them and ask about it, until it has completely resolved. The study sponsor may also ask the study doctor for this information.

   When the patient has completed the study, the doctor will then decide whether they require further treatment outside the study. They will continue to be followed up within the study every 8 weeks to document what other cancer treatment they may or may not be taking and to document overall survival. This contact may be in clinic if they are attending the hospital or can be by telephone if they are not.

   Timeline for Final Report The study is planned to recruit over 24 months with a further 12 months of follow up with final report planned for within 12 months of the last patient's last visit.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Female or male aged 18 years or older.
* Histologically proven metastatic or locally advanced inoperable squamous or adeno carcinoma of the oesophagus,stomach or oesophago-gastric junction.
* Documented progression after at least 1 prior line of chemotherapy for advanced disease. For HER2 positive tumours documented progression after at least 1 line of chemotherapy with or without HER2 directed therapy.
* c-MYC or HER2 gene amplification as defined in trial protocol
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study. If female patients are taking hormonal contraceptives to prevent pregnancy then this should be combined with a barrier method of contraception. Men must agree to not donate sperm during and after the study. For both males and females restrictions apply for 3 month after the last dose of study drug. See protocol for highly effective methods of birth control.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [b-hCG]) or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Mandatory provision of archival or fresh tumour biopsy for confirmation of c-MYC or HER2 gene amplification.
* World Health Organisation (ECOG) performance status 0-2, minimum life expectancy of 12 weeks from proposed first dose date, no deterioration within 2 weeks of screening and first dose.
* Adequate organ and haematological function as evidenced by the following laboratory values within 14 days before enrolment:

absolute neutrophil count (ANC) ≥1,500/mm3μL platelets ≥100,000/mm3μL (independent of transfusion support) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) total bilirubin ≤1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin serum creatinine ≤2 x ULN or estimated creatinine clearance (CCr) ≥30 mL/min/1.73m2

-At least one measurable target lesion, as per RECIST criteria 1.1

Exclusion Criteria:

* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Concurrent treatment within 4 weeks of study entry with any other chemotherapy, anticancer immunotherapy or experimental therapy
* No available histology for c-MYC or HER-2 amplification testing
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Patients with ECG abnormalities considered by the investigator to be clinically significant, or repeated baseline prolongation of the rate-corrected QT interval (QTc)
* Any actively bleeding gastrooesophageal tumour
* History of stroke or intracranial haemorrhage within 6 months prior to enrolment
* Symptomatic brain metastases
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
* Ongoing anticoagulation with a vitamin K antagonist
* Requiring use of strong P450 (CYP) 3A4 inhibitors
* Major surgery within 4 weeks of enrolment
* Vaccinated with live, attenuated vaccines within 4 weeks of enrolment
* Any pre-existing medical condition of sufficient severity to prevent full compliance with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2016-07-19 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate in patients with c-MYC and HER2 amplified advanced pre-treated oesophagogastric carcinomas treated with ibrutinib | 3 years
  Primary end point of objective overall radiological response rate, defined as confirmed complete response and partial response on CT or MRI imaging (assessed according to RECIST 1.1).

SECONDARY OUTCOMES:
Progression free survival | 3 years
  Defined as time from start of study treatment to disease progression or death from any cause. Will be analysed using the Kaplan-Meier method and the results presented as median survival with 95% confidence intervals.
Overall survival | 3 years
  defined as time from start of study treatment to death of any cause. Will be analysed using the Kaplan-Meier method and the results presented as median survival with 95% confidence intervals.
Disease control rate at 8 weeks | 8 weeks
  Proportion of patients with disease control (defined as complete response, partial response or stable disease by RECIST 1.1 on CT or MRI imaging) at 8 weeks.
Safety and tolerability of ibrutinib treatment in advanced oesophagogastric cancer | 3 years
  Assessing changes from baseline of laboratory data (clinical chemistry, haematology, urinalysis), vital signs & number of participants with adverse events (as assessed by CTCAE version 4)
Patient reported outcome- health related quality of life (HRQoL) as assessed by EORTC Quality of Life questionnaire QLQ-C30 | 3 years
  Quality of life subscale scores and change in subscale scores from baseline will be summarised separately by descriptive statistics (mean, median, standard deviation (SD), minimum, maximum) and presented graphically.
Patient reported outcome- health related quality of life (HRQoL) as assessed by EORTC Quality of Life questionnaire STO22 | 3 years
  Quality of life subscale scores and change in subscale scores from baseline will be summarised separately by descriptive statistics (mean, median, standard deviation (SD), minimum, maximum) and presented graphically.
Correlate metabolic changes on FDG-PET scan with changes in gene expression, circulating tumour cells and CT response | 3 years
  FDG-PET scan at baseline and day 14 will be correlated with changes seen in gene expression, circulating tumour cells and clinical response

OTHER OUTCOMES:
Pharmacokinetics of ibrutinib in advanced oesophagogastric cancer patients: Minimum Concentration (Cmin) of ibrutinib | 3 years
  Blood tests cycle 1 day 8 and cycle 1 day 14
Investigate dynamic changes in c-MYC copy number in circulating tumour DNA | 3 years
  Blood tests at pre screening, screening, cycle 1 day 14 and every 8 weeks whilst on treatment. Mandatory biopsy at screening, optional biopsies at day 14, disease response and progression
Correlate c-MYC amplification ratio in tumour tissue with c-MYC copy number variation in serum | 3 years
  Blood tests at pre screening, screening, cycle 1 day 14 and every 8 weeks whilst on treatment.Mandatory biopsy at screening, optional biopsies at day 14, disease response and progression

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chau, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Butler M, van Ingen Schenau DS, Yu J, Jenni S, Dobay MP, Hagelaar R, Vervoort BMT, Tee TM, Hoff FW, Meijerink JP, Kornblau SM, Bornhauser B, Bourquin JP, Kuiper RP, van der Meer LT, van Leeuwen FN. BTK inhibition sensitizes acute lymphoblastic leukemia to asparaginase by suppressing the amino acid response pathway. Blood. 2021 Dec 9;138(23):2383-2395. doi: 10.1182/blood.2021011787. PMID 34280258
- [Derived] Chong IY, Aronson L, Bryant H, Gulati A, Campbell J, Elliott R, Pettitt S, Wilkerson P, Lambros MB, Reis-Filho JS, Ramessur A, Davidson M, Chau I, Cunningham D, Ashworth A, Lord CJ. Mapping genetic vulnerabilities reveals BTK as a novel therapeutic target in oesophageal cancer. Gut. 2018 Oct;67(10):1780-1792. doi: 10.1136/gutjnl-2017-314408. Epub 2017 Aug 22. PMID 28830912